CLINICAL TRIAL: NCT02385708
Title: A Randomized Controlled Trial of 2% Chlorhexidine Gluconate Skin Preparation Cloths for the Prevention of Post-Operative Surgical Site Infections in Colorectal Patients
Brief Title: Use of 2% Chlorhexidine Cloths Reduce Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steven Klintworth, Research Nurse Specialist IV, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150309
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Patients will perform the current standard of care treatment using 2% Chlorohexidine Gluconate Cloths on the abdomen and buttocks prior to colorectal surgery night before surgery and morning of surgery
  Interventions: Drug: 2% Chlorohexidine Gluconate Standard of Care
- Treatment Arm (Active Comparator): Patients will perform treatment with 2% Chlorohexidine Gluconate cloths chin to toe night before and morning of surgery then daily post operative until post op day 4 or discharge
  Interventions: Drug: 2% Chlorohexidine Gluconate Chin to Toe

INTERVENTIONS:
Drug: 2% Chlorohexidine Gluconate Standard of Care — Patients will perform the current standard of care treatment using 2% Chlorohexidine Gluconate Cloths on the abdomen and buttocks prior to colorectal surgery night before surgery and morning of surgery.
  Other Names: 2% Chlorhexidine Gluconate
  Arms: Standard of Care
Drug: 2% Chlorohexidine Gluconate Chin to Toe — Patients will perform treatment with 2% Chlorohexidine Gluconate cloths chin to toe night before and morning of surgery then daily post operative until post op day 4 or discharge
  Other Names: 2% Chlorohexidine Gluconate
  Arms: Treatment Arm

SUMMARY:
Use of 2% chlorhexidine gluconate cloths pre-operatively and daily post-operatively jaw line to toes will decrease surgical site infections (SSI) by 30% when compared to patients who receive routine standard of care (use of chlorhexidine cloths night before surgery and morning of surgery).

DETAILED DESCRIPTION:
Patients undergoing colorectal surgery will be randomized in a 1:1 fashion into two groups. One will be standard of care using 2% Chlorhexidine Gluconate wipes night before surgery and morning if surgery. The second group will be randomized into the study arm using 2% Chlorhexidine Gluconate clothes from jaw line to toes night before surgery, morning of surgery and daily post operative. Skin cultures will be obtained at time of consent, prior to surgical procedure before surgical scrub and draping, post operative day 4 and at 30 day follow up visit. Incision lines will be assessed daily by study staff for signs of surgical site infection utilizing the CDC's 3 definitions of surgical site infections, superficial incisional SSI, deep incisional SSI, and organ space SSI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients > 18 years old scheduled for a colorectal surgical procedure ASA>2 OR pre-operatively hospitalized

Exclusion Criteria:

* Unable to consent
* Known allergy to any of the ingredients contained in SAGE chlorhexidine gluconate cloths
* Current infection or history of abdominal infections.
* Patients on chronic steroids or immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Klintworth, RN, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Fry DE. The prevention of surgical site infection in elective colon surgery. Scientifica (Cairo). 2013;2013:896297. doi: 10.1155/2013/896297. Epub 2013 Dec 19. PMID 24455434
- [Background] Grade M, Quintel M, Ghadimi BM. Standard perioperative management in gastrointestinal surgery. Langenbecks Arch Surg. 2011 Jun;396(5):591-606. doi: 10.1007/s00423-011-0782-y. Epub 2011 Mar 30. PMID 21448724
- [Background] Kobayashi M, Mohri Y, Inoue Y, Okita Y, Miki C, Kusunoki M. Continuous follow-up of surgical site infections for 30 days after colorectal surgery. World J Surg. 2008 Jun;32(6):1142-6. doi: 10.1007/s00268-008-9536-6. PMID 18338205
- [Background] Konishi T, Watanabe T, Kishimoto J, Nagawa H. Elective colon and rectal surgery differ in risk factors for wound infection: results of prospective surveillance. Ann Surg. 2006 Nov;244(5):758-63. doi: 10.1097/01.sla.0000219017.78611.49. PMID 17060769
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Surgical Site Infection: Prevention and Treatment of Surgical Site Infection. London: RCOG Press; 2008 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK53731/ PMID 21698848
- [Background] Smith RL, Bohl JK, McElearney ST, Friel CM, Barclay MM, Sawyer RG, Foley EF. Wound infection after elective colorectal resection. Ann Surg. 2004 May;239(5):599-605; discussion 605-7. doi: 10.1097/01.sla.0000124292.21605.99. PMID 15082963
- [Background] Stulberg JJ, Delaney CP, Neuhauser DV, Aron DC, Fu P, Koroukian SM. Adherence to surgical care improvement project measures and the association with postoperative infections. JAMA. 2010 Jun 23;303(24):2479-85. doi: 10.1001/jama.2010.841. PMID 20571014
- [Background] Watanabe M, Suzuki H, Nomura S, Maejima K, Chihara N, Komine O, Mizutani S, Yoshino M, Uchida E. Risk factors for surgical site infection in emergency colorectal surgery: a retrospective analysis. Surg Infect (Larchmt). 2014 Jun;15(3):256-61. doi: 10.1089/sur.2012.154. Epub 2014 May 8. PMID 24810804

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Patients will perform the current standard of care treatment using 2% Chlorohexidine Gluconate Cloths on the abdomen and buttocks prior to colorectal surgery night before surgery and morning of surgery
  2% Chlorohexidine Gluconate: Use of 2% Chlorhexidine cloths chin to toes daily
- Treatment Arm: Patients will receive detailed instruction for use of 2% Chlorohexidine Gluconate cloths chin to toe night before and morning of surgery then daily post operative till discharge
  2% Chlorohexidine Gluconate: Use of 2% Chlorhexidine cloths chin to toes daily
Period: Overall Study
Arm/Group | Standard of Care | Treatment Arm
Started | 81 | 82
Intervention Started | 81 | 82
Completed | 73 | 67
Not Completed | 8 | 15
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Withdrawn - surgery canceled | 2 | 5
Not completed — Investigator decision | 5 | 7
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Treatment Arm | Total
Number analyzed (Participants) | 73 | 67 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 39 | 87
  >=65 years | 25 | 28 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 47 | 43 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 72 | 67 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 1 | 9
  White | 65 | 66 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 67 | 140

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Surgical Site Infections
Description: Number of participants who had surgical site infection development at 30 day post operative visit based on Center for Disease Control Criteria for Defining A Surgical Site Infection (SSI), 2011.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Treatment Arm
Number analyzed (Participants) | 73 | 67
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From one day prior to surgery to post operative day 4
Arm/Group | Standard of Care | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/81 | 0/82
Other Adverse Events (participants affected / at risk) | 2/81 | 3/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=81) | Treatment Arm (N=82)
Anastomotic leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=81) | Treatment Arm (N=82)
Acute altered mental status change (Nervous system disorders) | 0 (0) | 1 (1) — resulting in escalation in level of care
nausea/vomiting/dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) — resulting in escalation in level of care
skin rash and itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
new onset atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0)
persistent tachycardia with hemodynamic instability (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02385708/Prot_SAP_000.pdf